CLINICAL TRIAL: NCT01920750
Title: Phase I Study to Evaluate New Leprosy Skin Test Antigens: MLSA-LAM and MLCwA
Brief Title: Leprosy Skin Test Antigens Phase 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 98-011
Record Dates: First submitted 2013-07-25; First posted 2013-08-12 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2013-08

CONDITIONS: Leprosy
Keywords: Leprosy, skin test, MLSA-LAM, MLCwA, diagnosis, Protocol 98-202
MeSH Terms: conditions — Leprosy; Disease

ARMS (2):
- Group 2 (Experimental): 5 subjects will receive d single 0.1 ml intracutaneous injections of 3 titrated doses (1, 10, and 25 grams/ml) of MLCwA and one of mock antigen equally in two arms
  Interventions: Biological: MLCwA; Biological: MLSA-LAM; Other: Mock Antigen
- Group 1 (Experimental): 5 subjects received single 0.1 ml intracutaneous injections of 3 titrated doses (1, 10, and 25 grams/ml) of MLSA-LAM and one of mock antigen equally in two arms
  Interventions: Biological: MLCwA; Biological: MLSA-LAM; Other: Mock Antigen

INTERVENTIONS:
Biological: MLCwA — Antigen MLSA-LAM is a pellet extracted 3x followed by removal of SDS by column chromatography. Contains many of the same proteins
Biological: MLSA-LAM — Antigen MLSA-LAM is derived from M. leprae extract following sonication and centrifugation, leaving the cytosol (MLSA). Contains soluble protein antigens of M. leprae
Other: Mock Antigen — Physiological saline

SUMMARY:
This is a small Phase I trial to evaluate the safety of the use as skin test antigens of the immunologically active proteins from the soluble/cytosol and insoluble cell wall of Mycobacterium leprae. The overall objective is to generate new leprosy skin-test antigens, equivalent to tuberculin-PPD in the tuberculosis context, to be used (I) for the early diagnosis of leprosy; and (ii) as epidemiological tools to measure the incidence of disease. Evaluating new leprosy skin test antigens may provide a better way to diagnose leprosy in its early stages of infection. With the early administration of drug therapy, infected individuals can then be cured of this disease before nerve damage occurs or nodules (lepromas) start to develop on the skin. Ten healthy, leprosy-unexposed, tuberculin-negative volunteers, 18-40 years old, from within the staff of the Mycobacteria Research Laboratories, Department of Microbiology, Colorado State University, Fort Collins, Colorado, will be selected.

DETAILED DESCRIPTION:
This is a small Phase I trial to evaluate the safety of the use as skin test antigens of the immunologically active proteins from the soluble/cytosol and insoluble cell wall of Mycobacterium leprae. The overall objective is to generate new leprosy skin-test antigens, equivalent to tuberculin-PPD in the tuberculosis context, to be used (I) for the early diagnosis of leprosy; and (ii) as epidemiological tools to measure the incidence of disease. Evaluating new leprosy skin test antigens may provide a better way to diagnose leprosy in its early stages of infection. With the early administration of drug therapy, infected individuals can then be cured of this disease before nerve damage occurs or nodules (lepromas) start to develop on the skin. Ten healthy, leprosy-unexposed, tuberculin-negative volunteers, ages 18-40 years old, from within the staff of the Mycobacteria Research Laboratories, Department of Microbiology, Colorado State University, Fort Collins, Colorado, will be selected for this study. The volunteers will be recruited by direct contact after placing notices in the Department of Microbiology at Colorado State University. There are approximately 40 faculty/staff/students in this population and all are routinely tested (PPD skin-testing or chest X-ray) by the staff at the Hartshorn Health Service Center in the context of the Department's tuberculosis research. Five individuals will be selected for testing MLSA-LAM and five will receive MLCwA. Each will receive single 0.1 ml intracutaneous injections of three titrated doses (1, 10 and 25 )lg/ml) of the skin-test antigen, one of mock antigen (i.e., physiological saline), and one of control antigen (the product now in use; Rees MLSA, 10 )lg), divided equally between the subject's two arms. Results will be recorded at 15 min, 48 h, 72 h, and 28 days post-injection. The test dose will be administered with a sterile1 ml syringe calibrated in tenths and fitted with a sterile, one-half inch, 26 or 27 gauge needle. The rubber stopper of the vial will be wiped with a sterile piece of cotton moistened with alcohol and allowed to dry.It is expected that all concentrations of the two leprosy skin test antigens will evoke similar negative responses. If so, all three concentrations will be used for subsequent studies. This protocol is linked to study 98-202.

ELIGIBILITY:
Inclusion Criteria:

* Born in the United States (less chance of previous exposure to tuberculosis or leprosy)
* Healthy individuals who are free of any evidence of leprosy or tuberculosis by established clinical examinations
* Between the ages of 18 and 40 years old
* Females of child-bearing age (defined from the period of menarche to menopause, usually between the ages of 15 to 45), certified as not pregnant (as determined by a pregnancy test performed within 7 days prior to admission into the study)
* Agreement to participate in the study after verbal explanation by the physician and nurses and signing of an informed consent form.
* Weight greater than 100 lbs. (female) and.140 lbs. (male)
* No known hypersensitivities or allergies
* Negative tuberculin skin test (as determined by skin tests performed 3 weeks prior to study entry)

Exclusion Criteria:

* Pregnant or lactating females
* Oral corticosteroid treatment
* Chronic illness
* Immunosuppressive condition
* Tuberculosis
* Leprosy
* Age <18 or >40
* Weight <100 lbs. (female) or <140 lbs. (male)
* Positive tuberculin skin test
* Extensive travel (2-3 trips/year) in leprosy/tuberculosis endemic regions

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 1989-01; Primary Completion 1999-02 (Actual); Study Completion 1999-02 (Actual)

PRIMARY OUTCOMES:
Range of concentration (1, 10, and 25 micrograms/ml) responses in the two leprosy skin test antigens in the control and mock antigens | Up to 28 days post injection
Incidence of leprosy | Up to 28 days post injection

REFERENCES:
- [Result] Rivoire BL, Groathouse NA, TerLouw S, Neupane KD, Ranjit C, Sapkota BR, Khadge S, Kunwar CB, Macdonald M, Hawksworth R, Thapa MB, Hagge DA, Tibbals M, Smith C, Dube T, She D, Wolff M, Zhou E, Makhene M, Mason R, Sizemore C, Brennan PJ. Safety and efficacy assessment of two new leprosy skin test antigens: randomized double blind clinical study. PLoS Negl Trop Dis. 2014 May 29;8(5):e2811. doi: 10.1371/journal.pntd.0002811. eCollection 2014. PMID 24874401